CLINICAL TRIAL: NCT01468714
Title: A Phase I, Open-Label, Fixed Sequence Study To Estimate The Steady-State Effect Of Ketoconazole On The Single-Dose Pharmacokinetics Of PF-04937319 In Healthy Adult Subjects
Brief Title: A Study To Estimate The Effect Of Ketoconazole On The Pharmacokinetics Of Pf-04937319 In Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: B1621011
Record Dates: First submitted 2011-10-04; First posted 2011-11-09 (Estimated); Last update posted 2011-11-16 (Estimated); Status verified 2011-11

CONDITIONS: Human Volunteers
Keywords: Drug Interaction; pharmacokinetics; ketoconazole; CYP3A
MeSH Terms: interventions — N,N-dimethyl-5-((2-methyl-6-((5-methylpyrazin-2-yl)carbamoyl)benzofuran-4-yl)oxy)pyrimidine-2-carboxamide; Ketoconazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: PF-04937319 / ketoconazole — Single 20 mg dose of PF-04937319 on day 1, multiple dose of ketoconazole 200 mg twice daily from day 3 to 7, single 20 mg dose of PF-04937319 on day 6

SUMMARY:
This study will evaluate the potential for a drug-drug interaction of PF-04937319 with ketoconazole, a potent inhibitor of the drug metabolizing enzyme CYP3A.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and/or female subjects between the ages of 18 and 55 years, inclusive. Healthy is defined as no clinically relevant abnormalities identified by a detailed medical history, full physical examination, including blood pressure and pulse rate measurement, 12-lead ECG or clinical laboratory tests.
* Body Mass Index (BMI) of 17.5 to 29.9 kg/m2; and a total body weight >=50 kg (110 lbs).
* Subjects of childbearing potential must agree to use a highly effective method of contraception throughout the study and for at least 28-days after the last dose of treatment.

Exclusion Criteria:

* Use of prescription or nonprescription drugs and dietary supplements within 7 days or 5 half-lives (whichever is longer) prior to the first dose of study medication.
* Pregnant or nursing females; females of childbearing potential who are unwilling or unable to use an acceptable method of non-hormonal contraception
* Consumption of grapefruit-containing products within 7 days prior to the first dose of study medication and while in the study protocol from at least 14 days prior to the first dose of study medication and for at least 28 days after the last dose of study medication

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2011-10; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Cmax of PF-04937319 | Day 1 & Day 6
Tmax of PF-04937319 | Day 1 & Day 6
AUClast of PF-04937319 | Day 1 & Day 6
(as data permits) AUCinf of PF-04937319 | Day 1 & Day 6
(as data permits) t1/2 of PF-04937319 | Day 1 & Day 6
Cmax of PF-04937319 M1 metabolite | Day 1 & Day 6
Tmax of PF-04937319 M1 metabolite | Day 1 & Day 6
AUClast of PF-04937319 M1 metabolite | Day 1 & Day 6
(as data permits) AUCinf of PF-04937319 M1 metabolite | Day 1 & Day 6
(as data permits) t1/2 of PF-04937319 M1 metabolite | Day 1 & Day 6

SECONDARY OUTCOMES:
Urinary recovery of PF-04937319 M1 metabolite | Day 1
(as data permits) renal clearance (CLr) of PF-04937319 M1 metabolite | Day 1

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, New Haven, Connecticut, United States

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B1621011&StudyName=A%20Study%20To%20Estimate%20The%20Effect%20Of%20Ketoconazole%20On%20The%20Pharmacokinetics%20Of%20Pf-04937319%20In%20Healthy%20Subjects